CLINICAL TRIAL: NCT02586662
Title: Prediction of Functional Disability in Subjects With Scapular Dyskinesis: Shoulder Tightness, Forward Shoulder Posture, Joint Range of Motion, Scapular Kinematics and Associated Muscular Activity
Brief Title: Prediction of Functional Disability in Subjects With Scapular Dyskinesis
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201112035RIB
Record Dates: First submitted 2015-10-14; First posted 2015-10-26 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Scapular Dyskinesis
Keywords: scapular dyskinesis; kinematics

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
Background: Patterns of scapular dyskinesis have unique scapular kinematics and associated muscular activation. The characteristics of scapular dyskinesis may be associated with functional disability. The investigators investigated whether the level of shoulder function and primary dysfunction items were different in each unique pattern of scapular dyskinesis. The factors associated with shoulder dysfunction in different patterns of scapular dyskinesis were identified.

Methods: Participants with unilateral shoulder pain were classified as having a single dyskinesis pattern (inferior angle prominence, pattern I; medial border prominence, pattern II) or a mixed dyskinesis pattern (patterns I+II). Clinical measurements with the Flexilevel Scale of Shoulder Function (FLEX-SF score), shoulder range of motion, anterior/posterior shoulder tightness, and pectoralis minor index were recorded. These clinical measurements, 3-D scapular kinematics (electromagnetic-based motion analysis), and associated muscular activation (electromyography on the upper, middle, and lower parts of the trapezius and serratus anterior muscles) during arm elevation were analyzed for associations with functional disability.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were from 18 to 50 years old and had unilateral shoulder pain around the shoulder complex, including the glenohumeral, scapulothoracic, sternoclavicular, and acromioclavicular regions, while performing shoulder movement.

Exclusion Criteria:

* Subjects were excluded if they had a history of shoulder dislocation, fracture, or shoulder surgery within the past 1 year, or a history of direct contact injury to the neck or upper extremities within the past 1 month. Subjects who had neurological disorders or demonstrated pain (VAS>3) during the overall testing procedures were also excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Function-related factors in patients with scapular dyskinesis. Fifty-one participants (40 males; 11 females; mean age= 22.5±2.4 years; mean height=171.4 ± 8.0 cm; mean weight= 64.9 ± 10.5 kg) were recruited.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Shoulder Function Questionnaire | one year
  Shoulder function of participants was assessed with the Flexilevel Scale of Shoulder Function (FLEX-SF score)
Range of Motion on shoulder, range in degrees | one year
  Shoulder range of motion of participants was assessed by a physiotherapist using goniometer to measure
Pectoralis Minor Index (PMI) | one year
  The length between the inferomedial aspect of the coracoid process and the caudal edge of the fourth rib at the sternum was measured by a physiotherapist using a meter, and then the parameter was divided by participants' height to calculate for PMI